CLINICAL TRIAL: NCT04324008
Title: Clinical Comparison of Different Flowable Resin Composites
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assistant Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flowable composites
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Tooth Diseases
Keywords: flowable resin composite; occlusal
MeSH Terms: conditions — Tooth Diseases; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Constic (Experimental): Constic (DMG, Hamburg, Germany)
  Interventions: Device: Constic
- G-ænial Universal Flo (Experimental): G-ænial Universal Flo (GC Corporation, Tokyo, Japan) in combination with G-Premio Bond (self-etch mode)
  Interventions: Device: G-ænial Universal Flo
- Tetric N-Flow (self-etch) (Experimental): Tetric N-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) in combination with Tetric N-Bond Universal (self-etch mode)
  Interventions: Device: Tetric N-Flow (self-etch)
- Tetric N-Flow (etch&rinse) (Experimental): Tetric N-Flow (Ivoclar Vivadent, Schaan, Liechtenstein) in combination with Tetric N-Bond Universal (etch&rinse mode)
  Interventions: Device: Tetric N-Flow (etch&rinse)

INTERVENTIONS:
Device: Constic — Flowable resin composite
  Arms: Constic
Device: G-ænial Universal Flo — Flowable resin composite
  Arms: G-ænial Universal Flo
Device: Tetric N-Flow (self-etch) — Tetric N-Flow (Tetric N-Bond Universal, self-etch mode)
  Arms: Tetric N-Flow (self-etch)
Device: Tetric N-Flow (etch&rinse) — Tetric N-Flow (Tetric N-Bond Universal, etch&rinse mode)
  Arms: Tetric N-Flow (etch&rinse)

SUMMARY:
The aim of this study is to evaluate a self-adhesive flowable resin composite, a flowable resin composite with high viscosity and a conventional flowable resin composite in combination with a universal adhesive using two different application modes. All patients will receive at least 4 occlusal restorations. Cavities will be divided into four groups according to restorative systems used: Constic (a self-adhering flowable composite), G-ænial Universal Flo (a highly filled flowable composite), Tetric N-Flow (self-etch) (a conventional flowable composite), Tetrin N-Flow (etch&rinse).

ELIGIBILITY:
Inclusion Criteria:

* having no medical or behavioral problems preventing then from attending review visits
* absence of previously placed restorations
* having antagonist teeth

Exclusion Criteria:

* poor gingival health
* uncontrolled, rampant caries
* bruxism
* removable partial dentures
* xerostomia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different flowable resin composite | two years
  Two year results according to USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)